CLINICAL TRIAL: NCT02434731
Title: Randomized Controlled Trial to Evaluate the Effectiveness of Vibration and External Cold (Buzzy Device) for Pain Relief During Venipuncture or Intravenous Cannulation in Children With Intellectual Disability.
Brief Title: Vibration and Cold for Pain Relief During Peripheral Intravenous Cannulation in Children With Intellectual Disability
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Principal Investigator, Ronfani Luca, MD, PhD, IRCCS Burlo Garofolo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC 20/13
Record Dates: First submitted 2015-04-27; First posted 2015-05-05 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Pain Relief
Keywords: Procedural pain; Phlebotomy; Intellectual Disability; Child; Buzzy
MeSH Terms: conditions — Pain, Procedural; Intellectual Disability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buzzy® device (Experimental): The Buzzy® device will be applied just above the selected site of the venipuncture; a ice pack will be attached under the device; the device will be turned on and after 15 second the procedure will be carried out.
  Interventions: Device: Buzzy® device
- No intervention (No Intervention): No intervention for pain relief

INTERVENTIONS:
Device: Buzzy® device — Buzzy® is a battery-powered device for venipuncture pain relief combining cold, vibration, and distraction.
  Arms: Buzzy® device

SUMMARY:
Needle procedures are the most common and important source of pain and distress in children in the health care setting. Children with intellectual disability from any cause experience pain more frequently than healthy children. They often require venipuncture or IV cannulation for diagnostic or therapeutic procedures. Pain in this population is often unrecognised because these patients are frequently unable to self-report their pain. Now it's possible to measure pain in children with intellectual disability with specific pain scales, like NCCPC-PV (Non-Communicating Children's Pain Checklist, Post-operative Version).

The efficacy of a device combining vibration and cold for pain relief during venipuncture or IV cannulation has been recently reported in children. The device's actions are based on the Gate Control Theory, whereby cold and vibrations stimulate large fiber and inhibitory neurons to interrupt nociception. This non-pharmacologic technique for pain relief could be useful in this kind of patients in emergency department. To date, there is no study that validated Buzzy device for pain relief in children with intellectual disability.

The aim of this study is to test the effectiveness of Buzzy® (a device that provides cold and vibration), in reducing the pain during venipuncture or IV cannulation, in children with intellectual disability.

ELIGIBILITY:
Inclusion Criteria:

* Age 4 to 17 years
* Presence of intellectual disability
* Need of peripheral IV line or venipuncture
* Informed consent signed by parents or legal guardians

Exclusion Criteria:

* Presence of abrasion, infection or break in skin in the area of Buzzy® placement
* Cold hypersensibility

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 71 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Pain score (NCCPC-PV scale) | intraoperative
  The pain during the procedure will be evaluated using the NCCPC-PV scale (Non-communicating Children's Pain Checklist - Postoperative Version) administered by a nurse

SECONDARY OUTCOMES:
Success at first attempt | intraoperative
  Percentage of success at first attempt
Number of attempts required | intraoperative
  Total number of attempts required
Adverse events | up to 15 minutes after the procedure
  The number and the type of adverse events will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Egidio Barbi, MD, Study Chair — IRCCS Burlo Garofolo, Trieste, Italy; Silvana Schreiber, RN, Study Director — IRCCS Burlo Garofolo, Trieste, Italy; Giorgio Cozzi, MD, Principal Investigator — IRCCS Burlo Garofolo, Trieste, Italy
Locations (1):
- IRCCS Burlo Garofolo, Trieste, Friuli Venezia Giulia, Italy

REFERENCES:
- [Derived] Schreiber S, Cozzi G, Rutigliano R, Assandro P, Tubaro M, Cortellazzo Wiel L, Ronfani L, Barbi E. Analgesia by cooling vibration during venipuncture in children with cognitive impairment. Acta Paediatr. 2016 Jan;105(1):e12-6. doi: 10.1111/apa.13224. Epub 2015 Nov 4. PMID 26401633